CLINICAL TRIAL: NCT04287504
Title: Validation of the OSOM BVBLUE Test for Bacterial Vaginosis and the SavvyCheck Vaginal Yeast Test for Vaginal Candidosis: A Prospective Study
Brief Title: Point-of-care Tests for Bacterial Vaginosis and Candidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alex Farr, MD PhD, Assistant Professor, Consultant Physician, Medical University of Vienna
Other Study IDs: 2115-2019
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Infection, Bacterial; Infection, Fungal; Preterm Birth
Keywords: point-of-care test; validation; preterm birth; bacterial vaginosis; candidosis
MeSH Terms: conditions — Bacterial Infections; Mycoses; Premature Birth; Vaginosis, Bacterial; Candidiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Yeast, control: Women negative for vulvovaginal candidosis on Gram stain smear.
  Interventions: Diagnostic Test: SavvyCheck Vaginal Yeast Test
- Yeast, study group: Women positive for vulvovaginal candidosis on Gram stain smear.
  Interventions: Diagnostic Test: SavvyCheck Vaginal Yeast Test
- Bacterial vaginosis, control: Women negative for bacterial vaginosis on Gram stain smear.
  Interventions: Diagnostic Test: OSOM BVBLUE Test
- Bacterial vaginosis, study group: Women positive for bacterial vaginosis on Gram stain smear.
  Interventions: Diagnostic Test: OSOM BVBLUE Test

INTERVENTIONS:
Diagnostic Test: SavvyCheck Vaginal Yeast Test — Point-of-care test for the detection of vaginal candidosis
  Groups: Yeast, control; Yeast, study group
Diagnostic Test: OSOM BVBLUE Test — Point-of-care test for the detection of bacterial vaginosis
  Groups: Bacterial vaginosis, control; Bacterial vaginosis, study group

SUMMARY:
Vaginal infection in early pregnancy is associated with an increased risk of spontaneous preterm delivery and late miscarriage. Most studies presume that vaginal infections are responsible for up to 40% of preterm birth. Although the causative microorganisms of vaginal infections are manifold, the three pathogens most commonly associated with vaginal infections are Gardnerella vaginalis, Candida albicans and Trichomonas vaginalis. The aim of this prospective study is the validation of the point-of-care tests OSOM BVBLUE for bacterial vaginosis and SavvyCheck Vaginal Yeast Test for candidosis in comparison to Gram stain.

DETAILED DESCRIPTION:
In the present study, it should be examined whether the OSOM BVBLUE for bacterial vaginosis and the SavvyCheck Vaginal Yeast Test for vaginal candidosis are superior, equal/comparable or inferior to diagnosis on Gram stained smears. The point-of-care-tests are potential tools for the adequate diagnosis of bacterial vaginosis and vaginal candidosis in early pregnancy, since the prevention of these infections, as well as the infection screening per se, have the potential to prevent preterm birth and reduce the rate of late abortion. Point-of-care-tests are easy to perform, relatively cheap, and widely available. Routine implementation of the tests would be an effective contribution to the reduction of preterm labor and late-onset mortality.

ELIGIBILITY:
Inclusion criteria:

* Legal age (Participants must be 18 years or over)
* Singleton pregnancy
* No recent therapy with antibiotics within the last two weeks
* No application of the following in the previous 72 hours before testing: vaginal ointments/crèmes, douches, spermicides, vaginal lubricants or feminine sprays

Exclusion criteria:

* Age below 18 years
* Multiple pregnancy
* Recent treatment with antibiotics
* Application of the following in the previous 72 hours: vaginal ointments/crèmes, douches, spermicides, vaginal lubricants or feminine sprays

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Study Population: Recruitement will take place during routine birth registration at the obstetric outpatient clinic at the Department of Obstetrics and Gynecology at the Medical University of Vienna. All data will be collected anonymized and encoded with numbers. Pregnant women will be screened for asymptomatic and symptomatic vaginal infection via Gram stain as part of routine management. Vaginal smears will be assessed by sterile swabs from the lateral vaginal wall and posterior fornix vaginae. Two swabs will be collected. The second swab will be taken for study purposes to undergo the OSOM BVBLUE Test for bacterial vaginosis or the SavvyCheck Vaginal Yeast Test for vaginal candidosis.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Test result of OSOM BVBLUE Test or SavvyCheck Vaginal Yeast Test | 10 minutes
  Result of point-of-care test

SECONDARY OUTCOMES:
Gestational age of delivery | approx. 6 months
  To assess preterm delivery rate

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kiss, MD MBA, Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dept. of Obstetrics and Gynecology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
on request